CLINICAL TRIAL: NCT06330987
Title: Recording and Study of Probable Fetal Electrocardiographic Signals From Maternal Electrocardiogram in Correlation With Fetal Autonomic Nervous sysTem Development.
Brief Title: Fetal Autonomic Nervous sysTem Evaluation
Acronym: FANTE
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Paolo Mannella, Full Professor of Obstetrics and Gynecology, University of Pisa
Other Study IDs: 15110_MANNELLA
Record Dates: First submitted 2024-02-29; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related; Pregnancy Disease; Pregnancy Complications; Pre-Eclampsia; Gestational Diabetes; ECG Electrode Site Reaction; Fetal Growth Retardation; Fetal Complications
Keywords: FANTE
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Diabetes, Gestational; Fetal Growth Retardation | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: electrocardiograph — Ten standard derivation electrodes were used to acquired FANTE registrations. The peripheral electrodes (Left (L), Right (R) and Foot (F)) were placed on the maternal abdomen in a triangle around the navel (orange) with lower apex, while the precordial ones (C1, C2, C3, C4, C5, C6) were put on an external circle. The Neutral electrode was on the right side of the patient abdomen. The software was configured so that the system acquired and wrote on disk 8 signals (2 bipolar and 6 referenced to the centroid of the three L, R and F leads) at 1000 sps with a resolution of 0.763uV. This high resolution is needed to resolve the very small voltage changes related to fetal cardiac activity.
  Other Names: Touch ECG HD+ (Cardioline S.p.A.)

SUMMARY:
The autonomic nervous system (ANS) is involved in cardiovascular, metabolic and cognitive processes, so its study in the fetus can provide relevant functional diagnostic and prognostic information. In particular, the study of the fetal ANS allows us to understand the degree of nervous maturation reached by the fetus and any developmental disorders that could have an impact on the cardiovascular characteristics of the fetus.

The goal of this open-label, non-randomized, prospective observational study is to study the fetal ANS in pregnant women between 23 and 40 weeks of gestation.

The objetives are:

* To Evaluate Fetal Autonomic Nervous System (FANTE) through the analysis of maternal electrocardiogram (ECG) and others clinical parameters usually used in pregnancy monitoring.
* To identify any variations in the fetal ECG in the event of developmental or pathological maternal and/or fetal pregnancy.

Participants will be recruited during ultrasound visits, information sessions, and hospitalizations after signing informed consent.

DETAILED DESCRIPTION:
The Autonomic Nervous System (ANS) is the main regulator of the body's homeostasis. It consists of two branches that work in balance: the sympathetic nervous system (SNS) and the parasympathetic nervous system (PNS). The SNS is responsible for the fight-or-flight response, while the PNS is responsible for the recovery response. The coordination of their actions is vital for the body's proper functioning. The two branches of the ANS develop asynchronously during fetal development, particularly from the vagus nerve (X pair of cranial nerves) within the PNS. However, its activity is severely limited by late myelination, and the tone of the SNP undergoes a first increase at around 25-32 weeks and a second increase at 37 weeks. In contrast, SNS maturation continues steadily throughout pregnancy. It has been recognized that imbalances in the development of the SNS may underlie intrauterine death, problems adapting to extrauterine life pediatric morbidity and increased risk of sudden infant death syndrome (SIDS). Altered ANS functioning has been linked to developmental pathologies in childhood, including autism spectrum disorders and other neuropsychiatric conditions, as well as adult cardiovascular and metabolic diseases. The causes of altered autonomic development are diverse, including factors related to pregnancy and pre-existing maternal pathologies. The primary causes are premature birth, abnormalities in placenta formation and development, intrauterine growth restriction (IUGR), maternal diabetes, hypothyroidism, substance abuse, and maternal mental illness.

Given this, evaluating the extent of ASN development may have significant implications not only in the obstetric and neonatal setting, but also in the long term. Sympathetic and parasympathetic tone indicators can be studied by examining Heart Rate Variability (HRV) on an electrocardiogram (ECG). Certain parameters can be detected in HRV that indicate different facets of autonomic tone, mainly the activity of the SNS (LF band), the PNS (HF band) and the sympathetic-vagal balance (LF/HF). Obtaining these parameters, however, requires the analysis of an electrocardiographic trace, which is not easy to acquire in intrauterine life.

The collaboration between the University of Pisa and the Institute of Clinical Physiology of the National Research Council of Italy (IFC-CNR) has led to the development of the FANTE method. FANTE (Fetal Autonomic Nervous Evaluation) enables the analysis of electrocardiographic traces acquired by placing electrodes on the maternal abdomen. The traces are interpreted using an algorithm developed by researchers at IFC-CNR, enabling extraction of HRV data with the same level of accuracy as fetal magnetocardiography. In sum, this method that allows accurate extraction of fetal ECGs from multichannel maternal abdominal signals. It represents a non-invasive and affordable option, which are fundamental characteristics for screening tools.

The assessment of FANTE has the potential to serve as a basis for risk stratification in populations affected by maternal or fetal disease. This tool may prove valuable for early diagnosis, allowing planning for more rigorous prenatal monitoring and comprehensive postnatal diagnosis.

Women with a singleton pregnancy attending or admitted to the Department of Obstetrics and Gynecology will be recruited between the 24th and 37th week of pregnancy. After signing the informed consent, they will be enrolled into the study.

At recruitment visit:

* Maternal anthropometric evaluation will be performed (age, body mass index (BMI), blood pressure smoking/alcohol/drug habits, medical therapies, or pathologies).
* Fetal well-being evaluation will be carried out by reviewing the reports of laboratory and ultrasound screening tests.
* The FANTE recordings will be performed using a 10-lead ECG placed on the maternal abdomen.

at FANTE periodic visit:

* FANTE registrations will be performed weekly.
* Standard maternal anthropometric assessments will be conducted as part of the periodic evaluations.

At delivery:

* Mode of delivery and any complications will be assessed.
* Within 48 hours of birth, anthropometric assessment of the infant according to clinical practice (weight, abdominal and head circumference).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy from 23 to 40 weeks of gestation.

Exclusion Criteria:

* Consent withdrawal
* Multiple pregnancy
* Singleton pregnancy below 23 weeks or above 40 weeks of gestation
* Contractions and signs of labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a singleton pregnancy attending or admitted to the Obstetrics and Gynecology Unit of the Santa Chiara Hospital, AOUP.
Sampling Method: Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Fetal Autonomic Nervous sysTem Evaluation (FANTE) | Between 23 and 40 weeks of pregnancy (Recording visit).
  The outcome measure assessed is heart rate variability (HRV), which is analyzed using the FANTE algorithm.
  HRV serves as an indicator of various facets of autonomic tone, including sympathetic (low frequency band, LF 0.04 - 0.15 Hz), parasympathetic (high frequency band, HF 0.15 - 0.4 Hz), and sympathetic-parasympathetic balance (LF/HF ratio) activity.
  Data are collected weekly, with each session lasting 10 minutes.

SECONDARY OUTCOMES:
Maternal Assesment | Between 23 and 37week of pregnancy (Recruitment visit).
  Occurrence of obesity, gestacional diabetes, habits such as smoking, alcohol, drug use, medical therapies, reports of maternal pathologies.
Obstetric Complications and mode of Delivery | Recruitment visit; Recording visit; Day of the delivery, in average 16 weeks after recruitment (post-partum visit).
  Occurrence of gestational hypertension, pre-eclampsia, intrauterine growth restriction, premature rupture of membranes, preterm labour.
  Mode of delivery (spontaneous, cesarean section, operative), neonatal weight and Apgar.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Mannella, MD. PhD., Principal Investigator — Department of Clinical and Experimental Medicine. University of Pisa
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No